CLINICAL TRIAL: NCT07106541
Title: Population Based Strategies for Standardized Surgical Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Anne Ehlers, Assistant Professor of Surgery, University of Michigan
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00278185
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Hernia, Abdominal
Keywords: Abdominal wall hernia repair; Surgical approach; Quality improvement in hernia care; Evidence-based guidelines; Replicating Effective Programs
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Intervention Model Description: Sites will get the REP package first. After this first stage of the SMART trial, non-responder MSQC-COHR hospitals (defined as hospitals that do not demonstrate ≥85% adherence to guidelines) will be randomized to continue REP versus REP with facilitation (REP-PLUS). The unit of randomization is the hospital. Stratified randomization on baseline site adherence will ensure comparability of comparators. In stage 2 non-responders in REP group will be re-randomized as well as the responders from the REP-PLUS group to REP vs REP-PLUS. The number of anticipated sites is listed as the anticipated enrollment numbers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Replicating Effective Programs (REP) - baseline program non-randomized (Experimental): All sites participating will be given this REP. This will be evaluated over 12 months.
  Interventions: Behavioral: Replicating Effective Programs (REP)
- REP with facilitation (REP-PLUS) - stage 1 randomized group (Experimental): Non-responders to the initial baseline program of REP MSQC-COHR hospitals (defined as hospitals that do not demonstrate ≥85% adherence to guidelines) randomized to this arm. This randomized arm will be evaluated over 12 months.
  Interventions: Behavioral: REP with facilitation (REP-PLUS)
- Replicating Effective Programs (REP) - stage 1 randomized group (Experimental): Non-responder to the initial baseline program of MSQC-COHR hospitals (defined as hospitals that do not demonstrate ≥85% adherence to guidelines) randomized to this arm. This randomized arm will be evaluated over 12 months.
  Interventions: Behavioral: Replicating Effective Programs (REP)
- Replicating Effective Programs (REP) (non-responders) - stage 2 randomized group (Experimental): Twelve months after the stage 1, non-responder MSQC-COHR hospitals (defined as hospitals that do not demonstrate ≥85% adherence to guidelines) that were assigned to the REP arm will be re-randomized to this arm or REP-PLUS. This randomized arm will be evaluated over 12 months.
  Interventions: Behavioral: Replicating Effective Programs (REP)
- REP with facilitation (REP-PLUS) (non-responders) - stage 2 randomized group (Experimental): Twelve months after the stage 1, non-responder MSQC-COHR hospitals (defined as hospitals that do not demonstrate ≥85% adherence to guidelines) that were assigned to the REP arm will be re- randomized to this arm REP-PLUS or REP alone. This randomized arm will be evaluated over 12 months.
  Interventions: Behavioral: REP with facilitation (REP-PLUS)
- REP-PLUS (responders) - stage 2 randomized group (Experimental): This group will include the REP-PLUS responders from stage 1. The responding hospitals will that are re-randomized to this group will continue to receive REP-PLUS.
  Interventions: Behavioral: REP with facilitation (REP-PLUS)
- Replicating Effective Programs (REP) (responders)- stage 2 randomized group (Experimental): This group will include the REP-PLUS responders from stage 1. The responding hospitals will that are re-randomized to this group will receive REP alone.
  Interventions: Behavioral: Replicating Effective Programs (REP)

INTERVENTIONS:
Behavioral: Replicating Effective Programs (REP) — The study team will deploy this stakeholder informed REP package across the 68 sites in the MSQC-COHR collaborative. The REP program uses a blend of formats including didactics, flipped classroom design, and narrative storytelling, the REP will address key barriers to adherence previously identified by surgeons.
  Arms: Replicating Effective Programs (REP) (non-responders) - stage 2 randomized group; Replicating Effective Programs (REP) (responders)- stage 2 randomized group; Replicating Effective Programs (REP) - baseline program non-randomized; Replicating Effective Programs (REP) - stage 1 randomized group
Behavioral: REP with facilitation (REP-PLUS) — This intervention is a stepped-up REP plus virtual facilitation. The facilitator will: 1) Initiate implementation and benchmark goals: The facilitator will partner with the identified site champions but be masked to primary and secondary outcomes. Together, the facilitator and site champions will review processes to organizationally embed clinical practice guidelines into practice, assess potential barriers and facilitators to these processes, and set measurable goals for adherence to recommendations; 2) Track adherence and provide feedback: Facilitators will use abstracted MSQC-COHR and site-specific operative data to track adherence to clinical practice guidelines, identify barriers to adherence, provide solutions to identified barriers, re-engage stakeholder groups responsible for unsatisfactory measurements, and continuously promote awareness of the guidelines.
  Arms: REP with facilitation (REP-PLUS) (non-responders) - stage 2 randomized group; REP with facilitation (REP-PLUS) - stage 1 randomized group; REP-PLUS (responders) - stage 2 randomized group

SUMMARY:
Evidence-based guidelines to improve clinical care for abdominal wall hernia repair are common, but adherence is low. This proposal aims to evaluate a stakeholder informed Replicating Effective Programs (REP) using a randomized controlled Sequential Multiple Assignment Randomized Trial (SMART).

The study team will leverage the 68-hospital Michigan Surgical Quality Collaborative Core Optimization Hernia Registry (MSQCCOHR), a statewide collaborative focused on quality improvement in hernia care. The study team will explore optimal remediation strategies for underperforming sites as well as opportunities to de-intensify interventions for responder sites.

ELIGIBILITY:
Inclusion Criteria:

- All hospitals that participate in MSQC-COHR will be eligible to participate in the trial

Exclusion:

- Institutes that are not in the MSQC-COHR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Adherence to clinical practice guidelines | 12, 24, 36 months
  Data will be reviewed from the MSQC-COHR. This is defined as the proportion of persons undergoing abdominal wall hernia that receive guideline concordant hernia care. The study team will define a "responder" as a site that has demonstrated ≥85% adherence to all three clinical practice guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Ehlers, MD, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan and other Michigan Surgical Quality Collaborative sites, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No